CLINICAL TRIAL: NCT01848184
Title: A Multicentre Prospective Study in Patients Undergoing Ventral Hernia Repair by Open Approach With Intraperitoneal Positioning Using Parietex™ Composite Ventral Patch - Panacea Study.
Brief Title: A Prospective Study in Patients Undergoing Primary Ventral Hernia Repair Using Parietex™ Composite Ventral Patch
Acronym: Panacea
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVPCOV0293
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-10

CONDITIONS: Hernia
Keywords: PARIETEX Composite Ventral Patch; PCO VP OR PCOVP; Primary ventral hernia repair; Panacea
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PARIETEX™ Composite Ventral Patch: PARIETEX™ Composite Ventral Patch for primary ventral hernia repair by open approach with intra-peritoneal positioning
  Interventions: Device: PARIETEX™ Composite Ventral Patch

INTERVENTIONS:
Device: PARIETEX™ Composite Ventral Patch — PARIETEX™ Composite Ventral Patch for ventral hernia repair

SUMMARY:
The objective of this study is to assess the recurrence rate following the use of PARIETEX™ Composite Ventral Patch in primary ventral hernia repair by open approach with intra-peritoneal positioning.

DETAILED DESCRIPTION:
Prospective, multicenter, multinational non-comparative study.

Primary Endpoint: Primary hernia recurrence* rate at 24 month follow-up. The evaluation of hernia recurrence will be performed during a physical examination and by ultrasonography.

Secondary Endpoints: Primary hernia recurrence* rate at 1, 6 and 12 month follow-up. The evaluation of hernia recurrence will be performed during a physical examination and confirmed by ultrasonography.

(*Recurrence is defined as a clinically manifested bulge or a protrusion exacerbated by a Valsalva maneuver.)

Safety Parameters:

Deep and superficial infection (A Surgical Site Infection (SSI) will be defined in the study according to the Centers for Disease Control and Prevention (CDC) criteria for diagnosis of SSI).

Pain / Chronic pain Other post-operative complications (complications related to visceral adhesions, Ileus, seroma, hematoma...) Analgesics consumption Risk factors (severity and treatment) Efficacy Parameters: Recurrence of primary ventral hernia Operative time Time of the mesh positioning Length of Hospital Stay Ease of use (Mesh handling and manipulability, comfort of use …) Return to daily activities/ work Patient satisfaction Patient comfort (Carolina's™ Comfort scale (CCS) - QoL questionnaire)

Visit Schedule:

Baseline visit (Preoperative) & Operative/Discharge visit

Post-Op:

Phone call Day 10

1 month 6 months 12 months 24 months

Duration: 12 months recruitment and 24 months follow-up Up to 12 sites in Europe and the United States will be included in this study

ELIGIBILITY:
Inclusion Criteria:

* All patients (adult ≥ 18 years) at participating centres undergoing primary ventral hernia repair with the device by open approach
* Signed informed consent form by the patient or the legally authorized representative
* Intraoperative inclusion criteria :Size of the defect: ≤ 4 cm

Exclusion Criteria:

* Emergency procedure
* Current participation in other trials
* History of previous hernia at the same location.
* Pregnant women: Women who are known or suspected to be pregnant, or who are planning to become pregnant during the study follow-up period
* Patient < 18 years
* BMI > 35
* ASA score ≥ 4
* The investigator determined that the patient will not be able to comply with the required follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for a primary ventral hernia repair with mesh by open approach (scheduled for non-emergent elective surgery with PCO VP) will be assessed for potential study participation (screening) and will be recorded in the patient log.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital Ghent (Belgium); Lars N Jørgensen, MD, Principal Investigator — Bispebjerg Hospital, University of Copenhagen (Denmark); Carl Doerhoff, MD, Principal Investigator — Surgicare of MO (United States); Steven Hopson, MD, Principal Investigator — Hernia Centers of Excellence, VA (United States); Eric KULLMAN, MD, Principal Investigator — Medicinskt Centrum i Linköping (Sweden); Marco G MUZI, MD, Principal Investigator — Department of Surgery, University Hospital Tor Vergata, Roma (Italy); Simon NIENHUIJS, MD, Principal Investigator — Catharina Ziekenhuis, EJ EINDHOVEN (The Netherlands); Filip E Muysoms, MD, Principal Investigator — Algemene Heelkunde, AZ Maria Middelares Ghent (Belgium); Tim Tollens, MD, Principal Investigator — Imelda Hospital, Bonheiden (Belgium); Karl Leblanc, MD, Principal Investigator — Our Lady of the Lake Regional Medical Center, LA (United States); Mark Schwartz, MD, Principal Investigator — Monmouth Medical Center, NJ (United States); Vic Velanovich, MD, Principal Investigator — University of South Florida (United States)
Locations (10):
- United States (5):
  - University of South Florida, Tampa, Florida
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Surgicare of Missouri, Jefferson City, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Hernia Centers of Excellence, Yorktown, Virginia
- Belgium (3):
  - General Surgery - Imelda Hospital, Bonheiden
  - Department of Surgery, Algemene Heelkunde AZ Maria Middelares Ghent, Ghent
  - Universitair Ziekenhuis Gent, Ghent
- Department of Surgery K, Bispebjerg Hospital, University of Copenhagen, Copenhagen, Denmark
- Dr. ERIC KULLMAN, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berrevoet F, Doerhoff C, Muysoms F, Hopson S, Muzi MG, Nienhuijs S, Kullman E, Tollens T, Schwartz M, Leblanc K, Velanovich V, Jorgensen LN. Open ventral hernia repair with a composite ventral patch - final results of a multicenter prospective study. BMC Surg. 2019 Jul 16;19(1):93. doi: 10.1186/s12893-019-0555-z. PMID 31311545

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PARIETEX™ Composite Ventral Patch
Started | 126
Completed | 100
Not Completed | 26

BASELINE CHARACTERISTICS:
Population: Consented and enrolled population 126 (100.0) Completed Study 100 (79.4) Discontinued early 26 (20.6)
Arm/Group | PARIETEX™ Composite Ventral Patch
Number analyzed (Participants) | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 107
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 87
Region of Enrollment [Number; unit: participants]
  Sweden | 15
  Belgium | 40
  United States | 33
  Denmark | 16
  Italy | 11
  Netherlands | 11

OUTCOME MEASURES:

1. Primary Outcome: Primary Hernia Recurrence Rate at 24 Month Follow-up.
Description: The number of participants with hernia recurrence at 24 months, assessed during a physical examination and by ultrasonography.
Time Frame: 24 month follow-up
Population: 101 patients returned for 24 month Follow-Up Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PARIETEX™ Composite Ventral Patch
Number analyzed (Participants) | 101
Participants | 3

2. Secondary Outcome: Recurrence Rate at 1, 6 and 12 Month Follow-up
Description: The number of participants with hernia recurrence at 1 month, 6 month and 12 month follow-up visit.
Time Frame: 1, 6 and 12 month follow-up.
Population: The number analyzed reflects the number of participants who returned for 1 month, 6 month and 12 month follow-up visits.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Undergoing Primary Ventral Hernia Repair: Patients undergoing primary ventral hernia repair using PARIETEX™ Composite Ventral Patch (PCO-VP)
Arm/Group | Patients Undergoing Primary Ventral Hernia Repair
Number analyzed (Participants) | 126
Participants
  1 month follow-up: number analyzed (Participants) | 122
  1 month follow-up | 0
  6 month follow-up: number analyzed (Participants) | 114
  6 month follow-up | 2
  12 month follow-up: number analyzed (Participants) | 111
  12 month follow-up | 3

3. Other Pre Specified Outcome: Pain Score at Baseline, Discharge, Day10, 1 Month, 6 Months, 12 Months & 24 Months
Description: Pain evaluation as determined by a 10-point pain intensity numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain). Scores reported at Baseline, Discharge, Day10, 1 Month, 6 Months, 12 Months & 24 Months
Time Frame: Various (Baseline, Discharge, Day10, 1 Month, 6 Months, 12 Months & 24 Months)
Population: The number analyzed includes participants who completed the NRS pain scale
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hernia Patients Receiving Surgery: Number of participants receiving surgery with PARIETEX™ Composite Ventral Patch for primary ventral hernia repair
Arm/Group | Hernia Patients Receiving Surgery
Number analyzed (Participants) | 126
units on a scale
  Baseline: number analyzed (Participants) | 120
  Baseline | 2.1 (2)
  Discharge: number analyzed (Participants) | 123
  Discharge | 2.9 (1.91)
  Day 10: number analyzed (Participants) | 125
  Day 10 | 1.5 (1.48)
  1 Month: number analyzed (Participants) | 123
  1 Month | 0.5 (0.74)
  6 Months: number analyzed (Participants) | 107
  6 Months | 0.4 (0.73)
  12 Months: number analyzed (Participants) | 111
  12 Months | 0.2 (0.4)
  24 Months: number analyzed (Participants) | 103
  24 Months | 0.1 (0.63)

4. Other Pre Specified Outcome: Summary of Risk Factors at Baseline
Description: Summary of Risk factors at Baseline. Risk factors include: Smoker, Obesity, Diabetes T1 & T2, Cancer, Cardiovascular disease, Hypertension, COPD, Chronic desease requiring analgesic or corticoid consumption
Time Frame: Baseline
Population: Number of patients with risk factors at baseline
Measure: Number; unit: participants
Groups:
- Hernia Patients Enrolled at Baseline: All patients enrolled at Baseline and assessed for risk factors
Arm/Group | Hernia Patients Enrolled at Baseline
Number analyzed (Participants) | 126
participants
  Smoker | 54
  Obesity (BMI>=30) | 43
  Diabetes Type 1 | 0
  Diabetes Type 2 | 10
  Cancer | 8
  Cardiovascular Disease | 19
  Hypertension | 36
  COPD | 9
  Chronic Disease-Analgesic Consumption | 4
  Chronic Disease-Corticoid consumption | 3

5. Other Pre Specified Outcome: Mesh Handling Ease of Use During Surgery
Description: Ease of use (mesh handling and comfort of use). Surgeons were asked if they were satisfied or completely satisfied, unsatisfied or completely dissatisfied
Time Frame: Per- operative
Population: Overal patients treated with PCO Ventral patch
Measure: Count of Participants; unit: Participants
Groups:
- Ease of Use: Ease of use (mesh handling and manipulability, comfort of use …)
Arm/Group | Ease of Use
Number analyzed (Participants) | 126
Participants
  Completely satisfied | 78
  Satisfied | 42
  Unsatisfied | 5
  Completely dissatisfied | 1

6. Other Pre Specified Outcome: Other Relevant Data: Operative Time
Description: Operative time during surgery for all patient receiving PCO ventral patch
Time Frame: Per- operative
Measure: Mean (Standard Deviation); unit: min
Groups:
- Operative Time: Operative time during surgery
Arm/Group | Operative Time
Number analyzed (Participants) | 124
min | 36.2 (15.57)

7. Other Pre Specified Outcome: Other Relevant Data: Time of Mesh Positioning
Description: The time of the mesh positioning during surgery
Time Frame: Per- operative
Measure: Mean (Standard Deviation); unit: min
Groups:
- Time Mesh Positioning: Time positioning of the mesh
Arm/Group | Time Mesh Positioning
Number analyzed (Participants) | 124
min | 8.1 (3.35)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | PARIETEX™ Composite Ventral Patch
All-Cause Mortality (participants affected / at risk) | 1/126
Serious Adverse Events (participants affected / at risk) | 21/126
Other Adverse Events (participants affected / at risk) | 41/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PARIETEX™ Composite Ventral Patch (N=126)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PARIETEX™ Composite Ventral Patch (N=126)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Local swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3)
Wound infection (Infections and infestations) | 2 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 26 (26)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes